CLINICAL TRIAL: NCT01799642
Title: Qualitative Descriptors of Dyspnea During Exercise in Cystic Fibrosis
Brief Title: Evaluating Sensations of Breathlessness in Patients With Cystic Fibrosis
Acronym: CF_Dyspnea
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H13-00262
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Lung; Disease; Cystic Fibrosis; Healthy
Keywords: dyspnea; exercise; cystic fibrosis; neuromechanical dissociation
MeSH Terms: conditions — Lung Diseases; Cystic Fibrosis; Dyspnea; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic Fibrosis Patients: Participants with Cystic Fibrosis
- Healthy Controls: Participants who do not have cystic fibrosis and are otherwise healthy.

SUMMARY:
Shortness of breath (dyspnea) during exercise is a major source of distress and is a commonly reported symptom in patients with cystic fibrosis (CF). Due to the investigators' poor understanding of how dyspnea develops, there are no treatments that consistently reduce dyspnea in this population. The investigators aim to acquire a more comprehensive understanding of the physiological mechanisms of exertional dyspnea in CF patients. This study will likely identify an important physiological mechanism of dyspnea in CF and may contribute to the development and use of effective treatments to reduce dyspnea in this population.

The central hypothesis is that the impaired tidal volume (VT) response during exercise in CF, in the setting of increased ventilatory demand will give rise to different qualitative descriptions of exertional dyspnea compared with healthy age and sex-matched controls. Specifically, CF patients will select "increased work and effort" as their dominant descriptor of dyspnea up to the VT inflection/plateau. Beyond this point, CF patient's dominant descriptor will become "unsatisfied inspiration." In contrast, healthy control participants will report "increased work and effort" throughout all phases of exercise and will not report "unsatisfied inspiration", even after the VT inflection/plateau.

DETAILED DESCRIPTION:
The purpose of this study is to determine if sensations of breathlessness (dyspnea) are qualitatively and quantitatively different in patients with cystic fibrosis (CF) compared to age and sex-matched healthy controls during exercise, and to determine if these differences can be explained by differences in the ventilatory response to exercise.

Understanding the progression of dyspnea during exercise will enable the investigators to better understand the pathophysiological mechanisms of this debilitating symptom in patients with CF. A more comprehensive understanding of the mechanisms underlying exertional dyspnea may ultimately lead to new therapeutic interventions (pharmacologic and non pharmacologic) that would positively impact exercise limitations in CF. A healthy control group will enable investigators to better identify the "normal" physiological and perceptual responses to exercise so that direct comparisons to patients with CF may be drawn.

Experimental Overview: Participants with CF and healthy control participants will report to the exercise laboratory for one visit. Informed consent, medical history screening, evaluation of chronic activity-related dyspnea and anthropometric measurements will firstly be obtained. Subjects will then be familiarized with the cycle ergometer, breathing apparatus and symptom scales. This will be followed by simple spirometry testing. After which participants will rest prior to a symptom limited incremental cycle exercise test. Detailed physiological and sensory measurements will be obtained during the familiarization and exercise test sessions. Data from the exercise test will address our hypotheses.

Study Participants: The study will include 40 participants in total. Of the 40 participants, 20 will be patients with CF and 20 will be healthy age and sex-matched controls.

Exercise Protocol: A symptom-limited incremental exercise test will be performed using an electronically braked cycle ergometer according to recommended guidelines. The test will consist of steady-state rest for 10 minutes, a 1 minute warm-up at 0 watts, and 20 watt stepwise increases in work rate every 2 minutes until symptom-limitation.

Measurements Familiarization Session: Participants and control participants will exercise on the cycle ergometer at a very low work rate (0W and 20W) for 2 minutes at each intensity in order to become familiarized with the cycle ergometer, breathing apparatus and symptom scales (see details below).

Pulmonary Function: Spirometry and maximum respiratory pressures, will be performed according to standard recommendations. A commercially available cardiopulmonary testing system (Vmax 229d with Autobox 6,200 DL; SensorMedics, Yorba Linda, CA) will be used, and all measurements will be expressed as percent of predicted normal values.

Dyspnea Evaluation: Dyspnea intensity (defined as "the sensation of laboured or difficult breathing") and perceived leg discomfort will be evaluated at rest, every minute during exercise, and at peak exercise using the modified 10-point Borg scale on all testing visits. Participants will be asked to describe their dyspnea during exercise prior to the intensity ratings and at end-exercise using the following 3 descriptors: (1) "my breathing requires more work and effort" (work and effort); (2) "I cannot get enough air in" (unsatisfied inspiration); (3) "I cannot get enough air out" (unsatisfied expiration). None to all 3 of the descriptors can be chosen at any one time. Upon exercise cessation, participants will be asked to verbalize their main reason(s) for stopping exercise (i.e., breathing discomfort, leg discomfort, combination of breathing and legs, or some other reason) and to select qualitative descriptors of breathlessness using an established questionnaire.

Cardio-respiratory Responses to Exercise: Standard cardio-respiratory measures will be recorded on a breath-by-breath basis and averaged over 30-second epochs, including minute ventilation (V'E), oxygen consumption (VO2), carbon dioxide production (CO2), partial pressure of end-tidal CO2, VT, and breathing frequency (Vmax 229d with Autobox 6,200 DL; SensorMedics, Yorba Linda, CA). Operating volumes (i.e., end-expiratory and end-inspiratory lung volumes) will be derived from dynamic inspiratory capacity (IC) manoeuvres as previously described. An indirect measure of neural respiratory drive will be obtained non-invasively using bi-polar surface electromyography (EMG) electrodes placed over the right parasternal intercostals and sternocleidomastoid as previously described. For safety purposes, electrocardiography will be monitored using a 12-lead electrocardiogram (ECG), blood pressure will be measured using a manual sphygmomanometer, and arterial oxygen saturation will be monitored using pulse oximetry. All exercise tests will be administered by experienced exercise physiologists. Tests involving patients with CF and healthy controls will be supervised by a physician. Exercise tests will be terminated based on established criteria as per American College of Sports Medicine guidelines.

Muscle oxygenation and hemodynamics: Muscle oxygenation will be noninvasively monitored using near infrared spectroscopy in all participants. A four-channel continuous-wave near-infrared spectroscope (Oxymon M III, Artinis Medical Systems, BV, The Netherlands) will be used to determine oxyhemoglobin, deoxyhemoglobin, and total hemoglobin by measuring light attenuation at 760 and 864 nm wavelengths, and analyzed using algorithms based on the modified Beer-Lambert law. This data will be used for descriptive exploratory purposes to examine the relationship between muscle oxygenation of the leg (vastus lateralis) and respiratory muscles (sternocleidomastoid, parasternal, and intercostals), and sensory responses to exercise in CF patients.

Computed Tomography Phenotyping: Existing chest computed tomography (CT) scans, obtained through routine clinical practice, will be used for descriptive exploratory purposes to examine the relationship between the extent of bronchiectasis vs. mucus plugging vs. air trapping (based on CF-specific CT scoring) on the physiological and sensory responses to exercise in patients with CF.

Inflection Point of the VT and V'E Relationship: VT data will be averaged over 30-second epochs and will be plotted against V'E at rest and throughout all exercise intensities for each individual participant. The point at which VT deviates from linearity and begins to plateau will be defined as the inflection point of the VT and V'E relationship. Two different observers will determine the inflection point for each participant during the incremental exercise test by examining individual Hey plots.

Statistical Analysis Data will be presented as means ± standard deviation (SD) unless otherwise specified. Between group comparisons (CF vs. healthy control) for descriptive characteristics, exercise responses, and Borg ratings at standardized evaluation points (20 watt increments, VT/minute ventilation (V'E) inflection, and peak) will be compared using unpaired t-tests with Bonferroni corrections where appropriate. Pearson correlation coefficients will be used to examine the association between measured variables: parasternals electromyography, breathing pattern, operational lung volumes, Borg ratings, and exercise variables. Reasons for stopping exercise and qualitative descriptors of dyspnea will be analyzed as frequency statistics and compared between control and CF participants using the Fisher's exact test at standardized 20 watt increments in work-rate, VT/V'E inflection, and peak exercise. A P-value less than 0.05 will be regarded as statistically significant. Statistical analysis of the data will be performed using Stata v11.2 (StataCorp, Texas, USA).

Sample Size and Power Calculation: Determining adequate sample size for qualitative descriptors of dyspnea in CF is difficult because limited data exists in this population. Therefore, the sample size in the present study is based on previous studies of dyspnea intensity ratings and the VT response in patients with chronic obstructive pulmonary disease during exercise. In these studies, statistically significant results were detected using a sample size of 16, under the assumptions: a SD of approximately 1.5 units, a difference of approximately 1.5 units found between the VT/V'E inflection point and peak exercise, a two-sided test, 80% power, and α = 0.05. Thus a sample size of 20 participants in the present study will likely have adequate power for the investigators' analyses.

ELIGIBILITY:
Inclusion Criteria:

* CF patients (confirmed based on abnormal sweat chloride testing and/or CF Transmembrane Conductance Regulator (CFTR) genotyping)
* Between the ages of 19 to 50 (inclusive)
* Stable clinical status (CF: no changes in therapy in the past 4 weeks)
* Forced Expiratory Volume in 1 second (FEV1.0) >40% predicted
* Body mass index greater than 18 or less than 30
* Currently non-smoking or a past smoking history of less than 20 pack-years
* Able to read and understand English

Exclusion Criteria:

* A disease other than CF that could contribute to dyspnea or exercise limitation
* Having either of the chronic infections Mycobacterium abscessus or Burkholderia cepacia complex
* Contraindications to clinical exercise testing
* Use of supplemental oxygen or desaturation less than 85% with exercise
* Diagnosis of pneumothorax in the past 4 weeks

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The CF patients will be recruited from the St. Paul's Hospital Adult CF Clinic. Healthy control participants will be recruited from the Vancouver area.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine if dyspnea is qualitatively and quantitatively different in patients with cystic fibrosis compared with age and sex-matched healthy controls during exercise | Parameters will be measured during the 1 visit.
  Included will be 20 patients with cystic fibrosis (CF) who have no other pulmonary or extra-pulmonary limitation to exercise, as well as 20 healthy age and sex-matched control participants. All participants (CF and control) will perform an incremental symptom-limited cardio-pulmonary exercise test while detailed cardio-respiratory responses, dyspnea responses, muscle oxygenation and muscle hemodynamic data are measured.

SECONDARY OUTCOMES:
To determine if the dyspnea responses can be explained by differences in the ventilatory response to exercise. | Parameters will be measured during the 1 visit.
  Included will be 20 patients with cystic fibrosis (CF) who have no other pulmonary or extra-pulmonary limitation to exercise, as well as 20 healthy age and sex-matched control participants. All participants (CF and control) will perform an incremental symptom-limited cardio-pulmonary exercise test while detailed cardio-respiratory responses, dyspnea responses, muscle oxygenation and muscle hemodynamic data are measured. The point at which the tidal volume deviates from linearity and begins to plateau will be defined as the inflection point of the tidal volume and minute ventilation relationship. Two different observers will determine the inflection point for each participant during the incremental exercise test by examining individual Hey plots.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — UBC James Hogg Research Centre
Locations (1):
- UBC James Hogg Research Centre, St. Paul's Hospital, Vancouver, British Columbia, Canada